CLINICAL TRIAL: NCT06721793
Title: The Impact of a Caffeinated Sports Drink on Performance
Acronym: NRG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Stavros Kavouras, Professor, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FP00041543; AWD00039989 (Other: ASU)
Record Dates: First submitted 2024-10-03; First posted 2024-12-06 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Dehydration; Dehydration Related to Exercise
Keywords: caffeine; sports drinks; hydration
MeSH Terms: conditions — Dehydration | interventions — Water

STUDY DESIGN:
Intervention Model Description: Counter balanced cross-over design trial with 4 arms differing only on the type of drink consumed during exercise.
  Each trial includes 2 hours of cycling in a warm environment (32ºC), followed by strength and cognitive assessments.
Who Masked: Participant
Masking Description: The type of drink ingested by the subjects will be labeled with a letter in a generic water bottle. During the trial with water a non-caloric, non-sodium-containing sweetener will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Water (Placebo Comparator): Water masked with non-caloric and no-sodium
  Interventions: Dietary Supplement: Water (Placebo)
- Carbohydrate electrolyte solution (Experimental): 2% carbohydrate solution with 1,020 mg/L of Sodium
  Interventions: Dietary Supplement: carbohydrate electrolyte drink
- no-sugar electrolyte solution (Experimental): 1% carbohydrate solution with 1,060 mg/L of Sodium
  Interventions: Dietary Supplement: no-sugar electrolyte drink
- Caffeinated carbohydrate electrolyte solution (Experimental): 1% carbohydrate solution with 1,000 mg/L of Sodium, and 200mg/L Caffeine
  Interventions: Dietary Supplement: Caffeinated Carbohydrate and electrolyte drink

INTERVENTIONS:
Dietary Supplement: carbohydrate electrolyte drink — 2% carbohydrate solution with 1,020 mg/L of Sodium
  Arms: Carbohydrate electrolyte solution
Dietary Supplement: no-sugar electrolyte drink — 1% carbohydrate solution with 1,060 mg/L of Sodium
  Arms: no-sugar electrolyte solution
Dietary Supplement: Caffeinated Carbohydrate and electrolyte drink — 2% carbohydrate solution with 1,000 mg/L of Sodium, and 200mg/L caffeine
  Arms: Caffeinated carbohydrate electrolyte solution
Dietary Supplement: Water (Placebo) — flavored water with non-caloric, non-sodium-containing sweetner
  Arms: Water

SUMMARY:
Caffeine is known to enhance physical and mental performance, but few beverages combine caffeine with electrolytes and carbohydrates to enhance exercise performance. This study evaluates a caffeinated electrolyte-glucose drink's effect on endurance, strength, and cognition. Using a repeated-measures, cross-over design, 20 trained cyclists will complete one familiarization and four randomized 3-hour experimental trials (Liquid I.V.™ Energy Multiplier, Hydration Multiplier, Sugar-Free Hydration Multiplier, and water). Each trial includes 2 hours of cycling in a warm environment (32ºC), followed by strength and cognitive assessments. Cycling performance, capillary blood, urine, and expiratory gases will be collected.

DETAILED DESCRIPTION:
Each subject will complete 5 trials (1 familiarization and 4 experimental) consisting of approximately 2 hours cycling in a warm environment (90ºF), followed by strength assessment and cognitive assessment via questionnaire. Each trial will be identical, with the only difference being the type of drink consumed during each trial. The first trial will be for familiarization without any blood sampling. The rest of the trials will be completed in a randomized order and the drink consumed

Cycling Endurance Exercise Performance

The exercise test will consist of a series of three consecutive cycling sets in a warm environment (90ºF), with each series consisting of:

1. a 30-min submaximal ride (50% maximal power as determined from the initial)
2. a 5-km time trial race-like performance effort. During each 30 min submaximal rides participants will drink a total 500 mL of fluid spread out during the 30 min. During the 5 km performance test the participants will drink 25 mL of fluid at the end of each kilometer.

At regular intervals throughout the exercise task, body weight, blood samples, respiratory gasses, and perceptual data will be collected. See study schematic provided below for specific measurement timepoints.

Upon completion of the cycling task subjects will moved to another room with cool temperature (70ºF), where strength and cognitive function will be assessed to determine the influence of each beverage on indices of exercise performance and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55
* Healthy and injury-free (muscle, skeletal) for greater than 2 months
* Active cyclists who train at least 3 times per week
* Body mass index (BMI) range of 18.5-30 kg/m2

Exclusion Criteria:

* • History of caffeine sensitivity

  * Cancer Diagnosis during the last 5 years
  * Pregnancy
  * History of renal disease, hypertension
  * History of a heat stroke
  * Use of testosterone therapy
  * Adults who are unable to consent (impaired decision-making capacity)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2025-12-12 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
5 kilometer cycling time trial | During the 3rd time trial which is the last time trial.
  Time in minutes of completion the 5 kilometer cycling time trial at the 3rd exercise bout.
5 kilometer Time trial performance | 2nd time trial
  Time to completion the 2nd cycling time trial
Isokinetic stregth | right after the cycling tests
  Peak torque at 60º/sec at dominant knee during extension
Congitive performance 1 | after the completion of strength test
  Attention Network Test score
Cognitive performance 2 | after the end of the strength assessment
  Working Memory Test score
Congitive test 3 | right after the strength test
  Stroop Task score

SECONDARY OUTCOMES:
Blood glucose | at the end of the 3rd cycling time trial.
  Blood glucose levels during the 3rd cycling time trial.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Kavouras, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University - Hydration Science Lab, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No